CLINICAL TRIAL: NCT07179367
Title: Innovative Teaching Method on the Patient Safety for Nursing Students: Escape Room
Brief Title: Escape Room for Patient Safety Training in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Demet SEMİZ, Lecturer, Fenerbahce University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24/286
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Patient Safety; Nursing Education
Keywords: Patient safety, escape room, nursing education, teaching methods

STUDY DESIGN:
Intervention Model Description: This study used a quasi-experimental, single-group pretest-posttest design. All participants received an escape room-based patient safety training, structured in three phases: prebriefing, simulation, and debriefing. Outcome measures were collected before and after the training.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- escape room training group (Experimental): This group consisted of fourth-year nursing students who received a patient safety-themed escape room training intervention. The simulation was structured in three phases: prebriefing, escape room activity, and debriefing. During prebriefing, students were oriented to the simulation environment and informed about patient safety principles. The escape room simulation consisted of three rooms designed according to INACSL standards, including scenarios on medication safety, maternal-infant care, and intensive care. Each room contained a mix of knowledge-based and skill-based tasks. After the simulation, a structured debriefing session was conducted using the PEARLS method to promote reflective learning. The intervention aimed to improve students' self-efficacy in patient safety practices and their satisfaction with the training method.
  Interventions: Other: Escape Room-Based Teaching Method on Patient Safety

INTERVENTIONS:
Other: Escape Room-Based Teaching Method on Patient Safety — Intervention Description: This intervention is a patient safety-themed escape room simulation specifically designed for nursing students. The activity consists of three phases structured in accordance with INACSL standards: pre-briefing, escape room simulation, and post-briefing assessment. Working in small groups, students solve knowledge- and skill-based patient safety tasks in three different rooms (patient safety, mother-baby room, and adult intensive care unit). Correct answers ensure progress, while post-briefing assessment using the PEARLS method supports reflection and learning. Unlike traditional teaching, this innovative method emphasizes teamwork, active participation, and experiential learning to increase self-efficacy and satisfaction with patient safety practices.

SUMMARY:
Ensuring patient safety is a cornerstone of nursing practice, and its foundation is established during nursing education. This study aims to empower senior nursing students to develop self-efficacy in patient safety practices through the "Escape Room" teaching method.

The study was conducted with senior nursing students from February to May 2024. Data were collected using the Student Information Form, Patient Safety Self-Efficacy Questionnaire, and Satisfaction with Training Methods Scale. The escape room was structured in three phases-prebriefing, simulation, and debriefing-following INACSL standards.

The average age of the participants was 23.5, and 43.5% had previously completed an elective course on patient safety. Analyses revealed that students spent the most time, averaging 2.59 minutes, in the room dedicated to information questions. The average self-efficacy score before the intervention was 61.26, which increased to 71.32 after the intervention, and participants reported a high level of satisfaction.

The study's findings indicate that patient safety-themed escape room training significantly enhances students' self-efficacy in patient safety, as well as their overall satisfaction and motivation.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Being a fourth-year nursing student at the Faculty of Nursing
* Completion of all data collection forms in full
* Volunteering to participate in the study

Exclusion Criteria:

* Staying in the escape room for more than 6 minutes in each room
* Not providing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Patient Safety Self-Efficacy | From baseline (pre-test, immediately before the escape room intervention) to post-test (immediately after the debriefing session, same day)."
  Primary Outcome Measure: Change in nursing students' patient safety self-efficacy scores from pre-test to post-test, measured by the Patient Safety Self-Efficacy Questionnaire (range: 0-75; higher scores indicate higher self-efficacy

SECONDARY OUTCOMES:
Satisfaction with Training Methods Scale | Immediately after completion of the escape room intervention (same day)
  Secondary Outcome Measure: Nursing students' satisfaction with the escape room training method, measured post-test by the Satisfaction with Training Methods Scale (range: 16-80; higher scores indicate higher satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Hamidiye Faculty of Nursing, University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT07179367/Prot_SAP_000.pdf